CLINICAL TRIAL: NCT02673502
Title: Impact of Pre-operative Carbohydrate Drink Provision on Attenuating Peri-operative Insulin Resistant in Major Abdominal Surgery: a Pilot Study
Brief Title: Pre-operative Carbohydrate Drink to Preserve Peri-operative Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Mitacs (Industry); Medtronic - MITG (Industry)
Responsible Party: Principal Investigator, Dr. Liane S. Feldman, Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-162-MUHC
Record Dates: First submitted 2016-01-28; First posted 2016-02-04 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Laparoscopic Abdominal Surgery
Keywords: Carbohydrate drink; Post operative complication; insulin resistance; Fasting blood glucose
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- simple carbohydrate drink (Experimental): Patients will ingest 400 ml of the simple carbohydrate drink consisting of commercial orange juice without pulp which contains 50 grams fructose/galactose 2 hours before surgery.
  Interventions: Dietary Supplement: simple carbohydrate drink
- complex carbohydrate drink (Experimental): Patients will ingest 400 ml of the complex carbohydrate drink containing 50 grams of maltodextrin powder in water ( orange food color and artificial orange flavor have been added to the drink) 2 hours before surgery.
  Interventions: Dietary Supplement: complex carbohydrate drink

INTERVENTIONS:
Dietary Supplement: simple carbohydrate drink — Patients will ingest 400 ml of the simple carbohydrate drink consisting of commercial orange juice without pulp which contains 50 grams fructose/galactose 2 hours before surgery.
  Arms: simple carbohydrate drink
Dietary Supplement: complex carbohydrate drink — Patients will ingest 400 ml of the complex carbohydrate drink containing 50 grams of maltodextrin powder in water ( orange food color and artificial orange flavor have been added to the drink) 2 hours before surgery
  Arms: complex carbohydrate drink

SUMMARY:
Enhanced Recovery after Surgery (ERAS) pathways include multiple evidence-based interventions delivered throughout the peri-operative period that aim to attenuate the surgical stress response and support rapid physiologic and functional recovery.A key element of the ERAS pathway is the administration of a clear carbohydrate-rich beverage 2-3 h before surgery in order to keep the patient in a fed state rather than a fasted state when they go to the operating room. The aim of the current study is to investigate the impact of a drink containing simple carbohydrate on attenuating surgical stress induced insulin resistance in patients undergoing major laparoscopic abdominal surgery, compared to drinks containing maltodextrin.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Planned laparoscopic partial colon resection for non-metastatic neoplastic or benign disease (including right, transverse, left or sigmoid))
3. HbA1c less than or equal to 5.7%
4. Not receiving any kind of glucose lowering medication.

Exclusion Criteria:

1. Are already diagnosed with diabetes or pre diabetes (HbA1c > 5.7%)
2. Are pre-diabetic receiving glucose lowering intervention (any glucose lowering medication)
3. Have renal or liver dysfunction (serum creatinine above 1.4 mg/dL in women and 1.5 mg/dL in men, bilirubin >2.9 mg/dL)
4. Will undergo extended resection of adjacent organs
5. Non-elective operations
6. New stoma created
7. Have conditions precluding participation in the ERAS pathway (e.g. dementia, disabling orthopedic and neuromuscular disease, psychosis)
8. Have conditions requiring preoperative fasting: documented gastroparesis, patient on metoclopramide and/or domperidone, achalasia, dysphagia (any difficulty with swallowing), or Fluid restriction (e.g. dialysis, pulmonary oedema, congestive heart failure).
9. Have cardiac abnormalities, severe end-organ disease such as cardiac failure (New York Heart Association classes III-IV), chronic obstructive pulmonary disease (documented by abnormal pulmonary function test), morbid obesity (BMI >40 kg/m2), anemia (hematocrit < 30 %, hemoglobin <100g/L, albumin < 25mg/dl)
10. Have received steroids for longer than 30 days
11. Have poor English or French comprehension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
difference in insulin resistance | Intra-operative from beginning of surgical procedure until the end of the procedure
  intra-operative insulin resistance as assessed by glucose infusion rate required to maintain euglycemic state during a hyperinsulinemic euglycemic glucose clamp

SECONDARY OUTCOMES:
Comparing the Homeostasis model assessment (HOMA) index at four different time points ( by employing Fasting blood sugar and Plasma Insulin) | at 4 time points as follow : on the morning before surgery, first, second and third morning after the surgery
Comparing the preoperative thirst | Two times at 2 weeks before surgery (baseline) and immediately before surgery
  Patients will complete a standard 10mm visual analogue scale (VAS) for each of the measures by marking the level on the scale at baseline in the pre-op clinic visit and once more immediately before surgery.
Comparing the preoperative hunger | Two times at 2 weeks before surgery (baseline) and immediately before surgery
  Patients will complete a standard 10mm visual analogue scale (VAS) for each of the measures by marking the level on the scale at baseline in the pre-op clinic visit and once more immediately before surgery.
Comparing the preoperative well-being | Two times at 2 weeks before surgery (baseline) and immediately before surgery
  Patients will complete a standard 10mm visual analogue scale (VAS) for each of the measures by marking the level on the scale at baseline in the pre-op clinic visit and once more immediately before surgery.
Comparing the preoperative anxiety | Two times at 2 weeks before surgery (baseline) and immediately before surgery
  Patients will complete a standard 10mm visual analogue scale (VAS) for each of the measures by marking the level on the scale at baseline in the pre-op clinic visit and once more immediately before surgery.
Grip strength | Two times at 2 weeks before surgery (baseline) and 2 days after surgery
  will be measured by a hand grip dynamometer
Time to readiness for discharge (TRD) | up to 30 days after surgery
  Previously described criteria to determine the time to readiness for discharge after colorectal surgery will be used . These criteria include tolerance of oral intake, recovery of lower gastro intestinal function, achieving adequate pain control, ability to mobilize and perform self-care and clinical/lab results showing no complications or untreated medical problems.
Postoperative infectious complications | 30 days after operation
  Including urinary tract infection, wound infection, intra- or retroperitoneal abscess, pneumonia , sepsis and any other documented infectious complications

CONTACTS AND LOCATIONS:
Overall Officials: Liane Feldman, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Francesco Carli, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada